CLINICAL TRIAL: NCT02804503
Title: The Effect of Menu Labels on Food Choices in Hispanics
Brief Title: The Effect of Menu Labels on Calories Ordered in Hispanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Meena Shah, Professor, Texas Christian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CT2016MS1
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Food Selection
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Calorie Labels (Experimental): A menu with rank ordered calorie labels and a statement on the energy needs per meal.
  Interventions: Behavioral: Calorie Labels
- Exercise Labels (Experimental): A menu with rank ordered exercise labels showing minutes of brisk walking necessary to burn the food calories.
  Interventions: Behavioral: Exercise Labels
- No Labels (Active Comparator): A menu with no labels
  Interventions: Behavioral: No Labels

INTERVENTIONS:
Behavioral: Calorie Labels — Participants were asked to order food from the assigned menu as if they were having lunch in a fast food restaurant.
  Arms: Calorie Labels
Behavioral: Exercise Labels — Participants were asked to order food from the assigned menu as if they were having lunch in a fast food restaurant.
  Arms: Exercise Labels
Behavioral: No Labels — Participants were asked to order food from the assigned menu as if they were having lunch in a fast food restaurant.
  Arms: No Labels

SUMMARY:
Most studies on menu labels have been conducted in mostly non-Hispanic white individuals, and how menu labels affect calories and macronutrients ordered in Hispanics is not clearly understood. This study evaluated the impact of menu labels on calories and macronutrients ordered in Hispanics.

DETAILED DESCRIPTION:
According to review studies, calorie labels on menus is not effective in reducing the number of calories ordered or consumed. Adding contextual information such as the energy needs per meal or interpretive information such as minutes of walking needed to burn the food calories or rank-ordering the food items from the lowest to the highest calorie content may be more effective in making food selections with fewer calories. Most studies on menu labels have, however, been conducted in mostly non-Hispanic white individuals, and how menu labels affect food choices in Hispanics in not well understood. This study evaluated the impact of menu labels on calories and macronutrients ordered in Hispanics by randomly assigning the participants to a menu with no labels (no labels), a menu with rank ordered calorie labels and a statement on the energy needs per meal (calorie labels), and a menu with rank ordered exercise labels (exercise labels). Calories and macronutrients ordered by the participants was assessed.

ELIGIBILITY:
Inclusion Criteria:

* Hispanics ages 18 through 65 years.

Exclusion Criteria:

* Not being able to read and write in either English or Spanish; pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Calories Ordered | 20-30 minutes
  Calories content of the food items ordered from the assigned menu was calculated.

SECONDARY OUTCOMES:
Macronutrients ordered | 20-30 minutes
  Macronutrients content of the food items ordered from the assigned menu was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Meena Shah, Ph.D., Principal Investigator — Tzu Chi University
Locations (1):
- Meena Shah, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Long MW, Tobias DK, Cradock AL, Batchelder H, Gortmaker SL. Systematic review and meta-analysis of the impact of restaurant menu calorie labeling. Am J Public Health. 2015 May;105(5):e11-24. doi: 10.2105/AJPH.2015.302570. Epub 2015 Mar 19. PMID 25790388
- [Result] Swartz JJ, Braxton D, Viera AJ. Calorie menu labeling on quick-service restaurant menus: an updated systematic review of the literature. Int J Behav Nutr Phys Act. 2011 Dec 8;8:135. doi: 10.1186/1479-5868-8-135. PMID 22152038
- [Result] Sinclair SE, Cooper M, Mansfield ED. The influence of menu labeling on calories selected or consumed: a systematic review and meta-analysis. J Acad Nutr Diet. 2014 Sep;114(9):1375-1388.e15. doi: 10.1016/j.jand.2014.05.014. Epub 2014 Jul 16. PMID 25037558
- [Derived] Shah M, Bouza B, Adams-Huet B, Jaffery M, Esposito P, Dart L. Effect of calorie or exercise labels on menus on calories and macronutrients ordered and calories from specific foods in Hispanic participants: a randomized study. J Investig Med. 2016 Dec;64(8):1261-1268. doi: 10.1136/jim-2016-000227. Epub 2016 Jul 8. PMID 27402619